CLINICAL TRIAL: NCT03309475
Title: Mindfulness-based Social Cognition Group Training (SocialMIND) Versus Psychoeducational Multicomponent Intervention in Patients With a First Episode of Psychosis (AGES-Mind Study): A Randomized Controlled Trial
Brief Title: Effectiveness of a Mindfulness-based Group Training Addressing Social Cognition in First Episode Psychosis (AGES-Mind)
Acronym: AGES-Mind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Carlos III Health Institute (Other Government); European Regional Development Fund (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGES-Mind
Record Dates: First submitted 2017-09-27; First posted 2017-10-13 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-10

CONDITIONS: Schizophrenia and Disorders With Psychotic Features; Psychotic Episode
Keywords: first episode psychosis; early psychosis; schizophrenia; mindfulness; social cognition; social functioning; AGES-Mind; SocialMind
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders; Psychotic Disorders; Schizophrenia; Social Adjustment

STUDY DESIGN:
Intervention Model Description: Pilot, multi-center, rater-blinded, prospective (48-weeks follow-up), randomized, controlled (versus active comparator [psychoeducation]), clinical trial. The experimental arm will receive treatment as usual (both drug and psychosocial therapy) and mindfulness-based social cognition group training, specifically designed for patients with first episode psychosis by the research team. The active comparator arm will receive treatment as usual (both drug and psychosocial therapy) and psychoeducation group training for psychosis.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The evaluators will not know the patients' assigned treatment arm until the end of the follow-up period. This information will only be delivered to investigators in charge of intervention groups, but not to those in charge of statistical analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SocialMIND (Experimental): The experimental arm will receive treatment as usual (both psychotropic treatment and psychosocial treatment) and mindfulness-based social cognition group training (SocialMind), specifically designed for patients with first episode psychosis by the research team. There will be a first phase (intensive intervention) consisting of 8 weekly sessions and a second phase (follow-up sessions) consisting of 4 fortnightly sessions and 5 monthly sessions.
  Interventions: Behavioral: SocialMIND; Behavioral: Psychosocial treatment; Drug: Psychotropic treatment
- Psychoeducational Multicomponent Intervention (Active Comparator): The active comparator arm will receive treatment as usual (both psychotropic treatment and psychosocial treatment) and a psychoeducational multicomponent intervention for psychosis.There will be a first phase (intensive intervention) consisting of 8 weekly sessions and a second phase (follow-up sessions) consisting of 4 fortnightly sessions and 7 monthly sessions.
  Interventions: Behavioral: Psychoeducational multicomponent intervention; Behavioral: Psychosocial treatment; Drug: Psychotropic treatment

INTERVENTIONS:
Behavioral: SocialMIND — SocialMind is a mindfulness-based intervention including elements such as radical acceptance, decentering or meditation-techniques. It is designed to target social cognition, defined as the ability to recognize, understand and benefit from social stimuli.
  Other Names: Mindfulness-based social cognition training; Mindfulness-based social cognition group training; MB-SCT
  Arms: SocialMIND
Behavioral: Psychoeducational multicomponent intervention — The psychoeducational multicomponent intervention addresses and discuss several aspects of great importance for persons who suffer a first episode of psychosis, such as biased perception and thinking, delusions-related anxiety or the nature of hallucinations. Its aim is to encourage patients to reflect upon their experiences from a critic perspective.
  Other Names: PMI; Structured psychoeducational group; Psychoeducational group; Psychoeducation group
  Arms: Psychoeducational Multicomponent Intervention
Behavioral: Psychosocial treatment — Treatment as usual delivered by patient's practitioner
Drug: Psychotropic treatment — Treatment as usual delivered by patient's practitioner
  Other Names: Drug treatment

SUMMARY:
The current investigation aims to compare two group intervention in patients with a first episode of psychosis, that is, people who have suffered their first psychotic episode within 5 years prior to their inclusion in the study. The experimental arm is a mindfulness-based social cognition training (SocialMind) designed by professionals with both formal training and clinical experience in the field of mindfulness and third generation cognitive-behavioral therapies. The active comparator arm is a psychoeducation program specifically designed for individuals with recent onset psychosis by members of the team with great experience in delivering such interventions. The main outcome is social functioning, as measured by the Personal and Social Performance Scale (PSP), an instrument developed for psychotic patients. The main hypothesis is that the improvement in social functioning will be larger among the participants on the experimental arm, because there is enough evidence suggesting that deficits in social cognition are present even in the first stages of psychotic syndrome and related to social functioning and general disability. Moreover, mindfulness-based interventions have proven themselves effective in other severe mental disorders.

DETAILED DESCRIPTION:
Social functioning is impaired among many patients with a first episode of psychosis, who also show a lower ability to recognize, understand and benefit from social stimuli (i.e., deficits in social cognition) than their pairs. Both deficits underlie the general functional impairment found across non-affective psychotic syndromes. Since currently available pharmacological strategies have not proven themselves effective in addressing this matter, new psychotherapeutic approaches should be developed. Investigators' main hypothesis is that a mindfulness-based social cognition group training (SocialMind) will improve social and general functioning, and that this improvement will be higher in the SocialMind than in the psychoeducation group. Given the association between oxidative stress and cognitive functioning, a relationship between oxidative stress biomarkers and intervention-related variables is also expected.

A research team with more than ten mental health professionals and many collaborators will carry and oversee the assessment sessions. A Pharmacology Department will analyse the biological samples. Regulated-trained, well-experienced clinicians will design and administer both interventions. The whole team will take part in the process of scientific publication and results dissemination.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* First hospitalization, first visit to mental health services with positive symptoms, onset of antipsychotic treatment, or first appearance of positive symptoms confirmed by an informant within the period of five years prior to the enrolment in the study;
* Informed consent given

Exclusion Criteria:

* Clinical Global Impression (CGI) higher than 5 ("markedly ill")
* Other Axis I diagnoses, except for substance use if psychotic symptoms remain at least 14 days after negative urine test.
* Intellectual disability plus impaired global functioning prior to disorder onset
* Generalized development disorder
* Pregnancy
* Attendance to either mindfulness programs or structured psychoeducational interventions at the time of the enrolment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in social functioning | 8, 16, 36 and 48 weeks
  Personal and Social Performance Scale (PSP) measures patient's functioning on different social areas, such as self-care, relationships, social activities and aggressive behavior.

SECONDARY OUTCOMES:
Change in global functioning | 8, 16, 36 and 48 weeks
  Global Assessment of Functioning Scale (GAF) measures patient's general functioning using a single 0-100 scale.
Change in quality of life | 8, 16, 36 and 48 weeks
  WHOQOL-BREF measures patient's quality of life according to World Health Organization parameters.
Change in clinical global impression | 8, 16, 36 and 48 weeks
  Clinical Global Impression Scale for Schizophrenia (CGI-SCH) measures patients' clinical state and clinical change over time
Change in psychotic symptoms | 8, 16, 36 and 48 weeks
  Positive and Negative Symptoms Scale for Schizophrenia (PANSS) measures psychotic syndrome through a detailed clinical interview.
Change in depressive symptoms | 8, 16, 36 and 48 weeks
  Calgary Depression Scale for Schizophrenia (CDSS) measures depressive symptoms in psychotic patients through a personal interview
Change in anxiety symptoms | 8, 16, 36 and 48 weeks
  Beck Anxiety Inventory (BAI) measures clinical anxiety through 21 items.
Change in social cognition | 8, 16, 36 and 48 weeks
  Hinting task, Reading the Mind in the Eyes Test (RMET), Emotion Recognition task (ER-40) and Ambiguous Intentions and Attribution Questionnaire (AIHQ) measure main domains of social cognition.
Change in reflective functioning | 8, 16, 36 and 48 weeks
  Reflective Functioning Questionnaire (RFQ-8) measures mentalization ability through a set of 8 questions
Change in emotional intelligence | 8, 16, 36 and 48 weeks
  Mayer-Salovey-Caruso Emotional Intelligence Test (MSCEIT v2.0) measures emotional intelligence through a set of questions referred to different situations.
Change in mindful attention and awareness | 8, 16, 36 and 48 weeks
  Mindfulness Attention Awareness Scale (MAAS) measures processes thought to be related to clinical outcomes in mindfulness-based interventions.
Change in cognitive insight | 8, 16, 36 and 48 weeks
  Beck Cognitive Insight Scale (BCIS) explores self-reflection and self-certainty, as parts of the cognitive insight construct
Change in neurocognition | 8, 16, 36 and 48 weeks
  Four tasks of the Matrics Consensus Cognitive Battery (MCCB) measure different domains of neurocognition (symbol coding, letter number span, spatial span and CPT-IP)
Change in oxidative stress and anti-inflammatory response | 8 and 48 weeks
  Total antioxidant status, enzymatic activity and cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Maria Fe Bravo, MD, PhD, Principal Investigator — Instituto para la Investigación Biomédica del Hospital universitario La Paz (IdiPAZ)
Locations (1):
- La Paz University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after the final results are published and for ever
Access Criteria: Researchers that are interested should contact the Principal Investigator

REFERENCES:
- [Background] Fond G, d'Albis MA, Jamain S, Tamouza R, Arango C, Fleischhacker WW, Glenthoj B, Leweke M, Lewis S, McGuire P, Meyer-Lindenberg A, Sommer IE, Winter-van Rossum I, Kapur S, Kahn RS, Rujescu D, Leboyer M. The promise of biological markers for treatment response in first-episode psychosis: a systematic review. Schizophr Bull. 2015 May;41(3):559-73. doi: 10.1093/schbul/sbv002. Epub 2015 Mar 10. PMID 25759473
- [Background] Brune M. "Theory of mind" in schizophrenia: a review of the literature. Schizophr Bull. 2005 Jan;31(1):21-42. doi: 10.1093/schbul/sbi002. Epub 2005 Feb 16. PMID 15888423
- [Background] Lecomte T, Corbiere M, Ehmann T, Addington J, Abdel-Baki A, Macewan B. Development and preliminary validation of the First Episode Social Functioning Scale for early psychosis. Psychiatry Res. 2014 May 30;216(3):412-7. doi: 10.1016/j.psychres.2014.01.044. Epub 2014 Feb 5. PMID 24613006
- [Derived] Mediavilla R, Munoz-Sanjose A, Rodriguez-Vega B, Bayon C, Palao A, Lahera G, Sanchez-Castro P, Roman E, Cebolla S, de Diego A, Pastor JM, Bravo-Ortiz MF. Mindfulness-based social cognition training (SocialMIND) versus psychoeducational multicomponent intervention for people with a first episode of psychosis: a study protocol for a randomised controlled trial. BMC Psychiatry. 2019 Jul 29;19(1):233. doi: 10.1186/s12888-019-2206-4. PMID 31357965
- See also: AGES-CM Consortium — http://www.agescm.es/index.php?lang=es